CLINICAL TRIAL: NCT00677261
Title: A Prospective, Unicenter, Randomized, Placebo Controlled, Clinical Interventional Trial, Comparing the Postoperative Functional Recovery as Well as Analgesic Efficacy of a Single Shot Sciatic Nerve Block Versus Posterior Capsule/Fat Pad Infiltration of Local Anesthetic for Total Knee Arthroplasty.
Brief Title: Comparing Postoperative Functional Recovery and Analgesic Efficacy of a Single Shot Sciatic Nerve Block Versus Posterior Capsule/Fat Pad Infiltration of Local Anesthetic for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Ben Safa, MD FRCPC Anesthesiologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 378-2007
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2011-07

CONDITIONS: Total Knee Arthroplasty; Post Operative Analgesia
Keywords: Knee; Arthroplasty; Sciatic; Nerve; Block; Regional; Anesthesia; Infiltration; Local Anesthetic; Analgesia
MeSH Terms: conditions — Bites and Stings; Agnosia | interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Procedure: Sciatic Nerve Block
- 2 (Experimental)
  Interventions: Procedure: Posterior capsule infiltration with local anesthetic
- 3 (Sham Comparator)
  Interventions: Procedure: Sham sciatic block and sham posterior infiltration

INTERVENTIONS:
Procedure: Sciatic Nerve Block — Patients randomized to Group 1 will receive a single sciatic nerve block using the infragluteal parabiceps approach, using 20 ml of 0.5 % Ropivacaine. A sham injection of the posterior capsule and fat pad using 50 cc of normal saline will be conducted at the conclusion of the surgery.
  Arms: 1
Procedure: Posterior capsule infiltration with local anesthetic — Patients randomized to Group 2 will receive a Sham sciatic nerve block using 20cc of normal saline as described above as well as extensive local anesthetic infiltration of the posterior capsule and fat pad with a solution of 50 ml of 0.2% ropivicaine.
  Arms: 2
Procedure: Sham sciatic block and sham posterior infiltration — Patients randomized to group 3 will only receive a continuous femoral nerve catheter, A sham sciatic nerve block with 20cc of normal saline as well as a sham injection of the posterior capsule and fat pad will be performed with 50cc of normal saline.
  Arms: 3

SUMMARY:
Many methods of pain relief have been implemented in an attempt to provide safe and effective analgesia for patients following total knee arthroplasty. Numerous studies have demonstrated that nerve blocks can provide superior pain control and reduce side effects. There are two major nerves that provide sensation to the knee: the femoral nerve provides sensation to the front of the knee and sciatic nerve provides sensation to the back of the knee. Putting local anesthetic close to these nerves provides superior pain control. The literature has supported the use of femoral nerve block for analgesia as well as improved functional outcome after total knee arthroplasty. The purpose of this study is to see if the same is true for sciatic nerve block for the back of the knee. We also would like to study an alternative approach to make the back of the knee pain free. This involves injecting local anesthetic directly into this area at the end of your surgery.Patients will be randomized into 3 groups: sciatic block, posterior infiltration of local anesthetic and placebo.This study will help further define the role of sciatic nerve block as well as the alternative technique of local anesthetic infiltration in the perioperative analgesic regimen of total knee arthroplasty surgery, in an effort to develop a standardized perioperative protocol for this patient population. The advent of this protocol should allow reduced risk, improved analgesia, and potentially earlier discharged from hospital with better function.

DETAILED DESCRIPTION:
The objectives of this study are:

1. Evaluate the role of sciatic nerve block in total knee replacement. There is conflicting data as to whether sciatic nerve block would provide significant analgesic benefit in addition to femoral nerve block and the usual multimodal and preemptive analgesic regimen for TKA.
2. Investigate the efficacy of single-shot sciatic nerve block on early rehabilitation, functional recovery and patient satisfaction.
3. Evaluate the previously described technique of local anesthetic infiltration into the posterior capsule/fat pad of the knee as an alternative technique to sciatic nerve block in providing analgesia to the posterior aspect of the knee in this select group of patients.
4. Investigate the efficacy of local anesthetic infiltration into the posterior capsule/fat pad of the knee on early rehabilitation, functional recovery and patient satisfaction.

Study Design:

All patients will have a femoral nerve block (FNB) and spinal anesthesia.

Patients will be randomized into one of the 3 possible groups:

Group 1: Femoral nerve block + Sciatic nerve block + Spinal anesthesia + Infiltration of normal saline at the end of surgery

Group 2: Femoral nerve block + Sham Sciatic nerve block + Spinal anesthesia + Infiltration of local anesthetic at the end of surgery.

Group 3: Femoral nerve block + Sham Sciatic nerve block + Spinal anesthesia. + Infiltration of normal saline at the end of surgery.

In summary, this study will help further define the role of sciatic nerve block as well as the alternative technique of local anesthetic infiltration in the perioperative analgesic regimen of total knee arthroplasty surgery, in an effort to develop a standardized perioperative protocol for this patient population. The advent of this protocol should allow reduced risk, improved analgesia, and potentially earlier discharged from hospital with better function.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I and III
* Scheduled for total knee arthroplasty

Exclusion Criteria:

* Patients not providing informed consent.
* Refusal of treatment plan.
* Preexisting medical/neurological/hematologic conditions contraindicated for spinal anesthesia or peripheral nerve blocks.
* Revision total knee arthroplasty.
* Known allergy to any of the medications being used.
* History of drug or alcohol abuse.
* Patients with chronic pain on slow-release preparations of opioid in excess of 30mg of morphine equivalence per day.
* Patients with Rheumatoid Arthritis.
* Patients with psychiatric disorders.
* Patients unable or unwilling to use Patient Controlled Analgesia.
* Diabetic patients or those with impaired renal function (Creatinine >106).
* Obese patients (i.e. BMI >45).
* Postoperatively, patients will be excluded if they have had additional operative procedures requiring a change in the usual rehabilitation protocol of care.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-06; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for pain will be used (0=no pain, 100mm = terrible pain) as our primary outcome, for 72 hours post-operatively (at rest and during mobilization). | On arrival to PACU and every 4 hours thereafter.

SECONDARY OUTCOMES:
The TUG (Timed up and go test) and Range of motion. | Performed on day 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Safa, MD, FRCPC, Principal Investigator — Staff Anesthesiologist, Sunnybrook Health Sciences Centre.
Locations (1):
- Holland Orthopedic and Arthritic Centre, Toronto, Ontario, Canada